CLINICAL TRIAL: NCT03859934
Title: Metabolic Effects of Melatonin Treatment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2019-000213-37
Record Dates: First submitted 2019-02-18; First posted 2019-03-01 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Metabolic Disease; Insulin Sensitivity; Glucose Metabolism Disorders (Including Diabetes Mellitus); Type 2 Diabetes Mellitus; Blood Pressure; Inflammation
MeSH Terms: conditions — Metabolic Diseases; Insulin Resistance; Glucose Metabolism Disorders; Diabetes Mellitus, Type 2; Inflammation | interventions — Melatonin

STUDY DESIGN:
Intervention Model Description: Randomized, placebo controlled, double blinded crossover study
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Melatonin (Active Comparator): 10 mg melatonin each day 1 hour before bedtime for 3 months
  Interventions: Drug: Melatonin
- Placebo (Placebo Comparator): Placebo each day 1 hour before bedtime for 3 months
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Melatonin — Melatonin treatment
  Other Names: Melatonin treatment
  Arms: Melatonin
Drug: Placebo Oral Tablet — Placebo treatment
  Other Names: Placebo treatment
  Arms: Placebo

SUMMARY:
Modern living is associated with an epidemic of type 2 diabetes mellitus (T2DM). Sleep disturbances such as insomnia or frequent awakenings are strong risk factors for T2DM with several studies indicating a central role of melatonin. Additionally, a certain single nucleotide polymorphism in the melatonin receptor gene, MTNR1B rs10830963, with an allele frequency of 30 %, is associated with increased fasting plasma glucose and T2DM. Due to treatment of, among other things, insomnia, the use of melatonin is increasing rapidly in Denmark with a 100-fold increase from 2007-2012 in children and adolescents. No previous studies have thoroughly assessed changes in glucose and fatty acid metabolism after 3 months of melatonin treatment in patients with T2DM.

DETAILED DESCRIPTION:
Modern living is associated with an epidemic of type 2 diabetes mellitus (T2DM). Sleep disturbances such as insomnia or frequent awakenings are strong risk factors for T2DM with several studies indicating a central role of melatonin. Additionally, a certain single nucleotide polymorphism in the melatonin receptor gene, MTNR1B rs10830963, with an allele frequency of 30 %, is associated with increased fasting plasma glucose and T2DM. Due to treatment of, among other things, insomnia, the use of melatonin is increasing rapidly in Denmark with a 100-fold increase from 2007-2012 in children and adolescents. No previous studies have thoroughly assessed changes in glucose and fatty acid metabolism after 3 months of melatonin treatment in patients with T2DM.

Main research questions:

1. Does chronic melatonin treatment change insulin secretion in T2DM patients?
2. Does chronic melatonin treatment change insulin sensitivity in T2DM patients?
3. Does the MTNR1B rs10830963 risk allele alter the insulin secretion and insulin sensitivity compared with carries of the normal variant after chronic melatonin treatment?
4. Does chronic melatonin treatment change insulin signalling in muscle - and adipose tissue? Design: A randomized, double-blinded, placebo controlled, crossover study, including 18 participants with T2DM. We aim to recruit 9 homozygous carriers of the normal allele and 9 hetero - or homozygous for the risk allele.

Participants will be examined on two occasions, 1) after 3 months of daily melatonin treatment before bedtime (10 mg), and 2) after 3 months of daily placebo treatment before bedtime.

On the study days, participants will initially undergo a basal period with glucose - and palmitate tracer infusions to assess endogenous glucose production and free fatty acid production. Afterwards a Botnia clamp, which combines an intravenous glucose tolerance test and a hyperinsulinemic euglycemic clamp, will be performed to assess β-cell function and insulin sensitivity. On both study days muscle - and fat biopsies will be performed under both basal and hyperinsulinemic euglycemic conditions.

Perspectives: It is highly relevant to evaluate the chronic effects of melatonin on glucose - and fat metabolism given the increase in melatonin consumption. Furthermore, the study may open for new treatment options of T2DM if beneficial effects of oral melatonin are detected.

ELIGIBILITY:
Inclusion Criteria:

* Male sex
* Caucasian race
* Type 2 Diabetes Mellitus (T2DM)
* T2DM duration of maximum 20 years
* Age 40-70 years
* BMI between 25-35 kg/m2 at T2DM debut
* Written consent prior to study participation

Exclusion Criteria:

* > 3 daily antihypertensive drugs
* Blood pressure > 160/100 mmHg
* Insulin treatment
* > 3 daily oral antidiabetic drugs
* > 1 lipid lowering drug
* HbA1c > 65
* Heart failure (New York Heart Association Class III or IV), liver disease (alanine aminotransferase (ALAT) > twice the upper limit of normal serum concentration), plasma creatinine > 130 µmol/L and/or albuminuria, goiter, active cancer, acute or chronic pancreatitis
* Treatment with antidiabetic medicine that cannot be paused on study days (or for a week if the participants is treated with longtime-acting GLP-1 analogs)
* Shift work within the last year
* Travel across >4 time zones planned within the next 6 months
* Use of melatonin on a regular basis within the last year
* Severe illness
* > 14 units of alcohol/week
* Previous diagnosis of a sleep disorder
* Present or earlier alcohol or drug abuse
* Unable to give informed consent
* Allergy towards melatonin
* Daily consumption of benzodiazepines, fluvoxamine, amiodarone, efavirenz, fluoroquinolones, rifampicin, and carbamazepine due to interactions with the pharmacokinetics of melatonin.
* Severe sleep apnea (>30 respiration breaks/hour over 10 seconds)
* Medical treated depression or anxiety disorders within the last 3 years
* Daily consumption of selective serotonin reuptake inhibitors or tricyclic antidepressants

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 17 (Actual)
Dates: Start 2019-09-26 (Actual); Primary Completion 2021-05-03 (Actual); Study Completion 2021-08-18 (Actual)

PRIMARY OUTCOMES:
Change of insulin sensitivity | The outcome will be measured after 3 months of placebo treatment and after 3 months of melatonin treatment and compared afterwards with a paired T-tes
  Insulin sensitivity is assessed by a hyperinsulinemic euglycemic clamp, unit: mg/kg/min (mg of glucose to maintain euglycemia per kilogram of weight per minuts)
Change of insulin secretion change | The outcome will be measured after 3 months of placebo treatment and after 3 months of melatonin treatment
  Insulin secretion is assessed by an intravenous glucose tolerance test, unit: pmol/L (insulin)
MTNR1a rs10830963 influence on change in insulin sensitivity and insulin secretion | The outcome will be measured after 3 months of placebo treatment and again after 3 months of melatonin treatment
  MTNR1a rs10830963 genotype influence on insulin sensitivity and insulin secretion (see outcome 1 + 2)
Change of insulin signalling | The outcome will be measured after 3 months of placebo treatment and after 3 months of melatonin treatment
  Insulin signalling in muscle and adipose tissue assessed by western blot

SECONDARY OUTCOMES:
Change of ambulatory blood pressure | The outcome will be measured after 3 months of placebo treatment and after 3 months of melatonin treatment
  Ambulatory blood pressure assessed with Mobil-O-graph, I.E.M., Stolberg, Germany (Unit: mmHg)
Change of arterial stiffness | The outcome will be measured after 3 months of placebo treatment and after 3 months of melatonin treatment
  Arterial stiffness assessed with Mobil-O-graph, I.E.M., Stolberg, Germany (unit: m/s)
Change of gut microbiome | The outcome will be measured after 3 months of placebo treatment and after 3 months of melatonin treatment
  Feces analysis of microbial mRNA
Change of sleep evaluation 1 | The outcome will be measured after 3 months of placebo treatment and after 3 months of melatonin treatment
  Pittsburg Sleep Quality Index Questionnaire (Points on a scale: range 0-57)
Change of sleep evaluation 2 | After 3 months treatmentThe outcome will be measured after 3 months of placebo treatment and after 3 months of melatonin treatment
  Epworth Sleepiness Scale Questionnaire (Points on a scale: range 0-24)
Change of psychological health 1 | The outcome will be measured after 3 months of placebo treatment and after 3 months of melatonin treatment
  Major Depression Inventory Questionnaires (points on a scale: range 0-65)
Change of psychological health 2 | The outcome will be measured after 3 months of placebo treatment and after 3 months of melatonin treatment
  World Health Organization 5 Questionnaires (points on a scale: range 0-25)
Hormonal changes | The outcome will be measured after 3 months of placebo treatment and after 3 months of melatonin treatment
  Ghrelin, HbA1c, GLP-1, GLP-2, GIP, free fatty acids (FFA), leptin, cytokines, adiponectin, growth hormone, cortisol, hsCRP, CD163, MBL, IGF-1 and proinsulin measured by ELISA, RIA, or routine biochemical analysis. Unit: pmol/L
Change of glucose and palmitate kinetics | The outcome will be measured after 3 months of placebo treatment and after 3 months of melatonin treatment
  Tracer technique with infusion of radioactive labeled glucose and palmitate for determination of rate of appereance. Unit: mikromol/min
Change of regional glucose and palmitate uptake | The outcome will be measured after 3 months of placebo treatment and after 3 months of melatonin treatment
  Forearm model with arteriovenous differences of glucose and palmitate (Arterial glucose minus venous glucose = forearm uptake (unit mmol/l). The same applies for palmitate
Change of DEXA-scans | The outcome will be measured after 3 months of placebo treatment and after 3 months of melatonin treatment
  Evaluation of body composition and bone mineral density by DEXA-scan
Change of assessment of respiratory quotient (RQ) | The outcome will be measured after 3 months of placebo treatment and after 3 months of melatonin treatment
  Assessment of respiratory quotient (RQ) with indirect calorimetry (unit: VCO2/VO2)
Change of assessment of resting energy expenditure (REE) | The outcome will be measured after 3 months of placebo treatment and after 3 months of melatonin treatment
  Assessment of resting energy expenditure (REE) with indirect calorimetry (Unit J/s)

CONTACTS AND LOCATIONS:
Overall Officials: Esben Stistrup Lauritzen, MD, Principal Investigator — Medical Research Laboratory; Ulla Kampmann Opstrup, MD, PhD, Principal Investigator — Aarhus University Hospital; Julie Støy, MD, PhD, Principal Investigator — Aarhus University Hospital
Locations (1):
- Medical Research Laboratory, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No